CLINICAL TRIAL: NCT05509933
Title: Budesonide Prophylaxis for Engraftment Syndrome After Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, MD, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15795
Record Dates: First submitted 2022-08-19; First posted 2022-08-22 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Engraftment Syndrome
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Budesonide (Experimental)
  Interventions: Drug: Budesonide
- nothing (No Intervention)

INTERVENTIONS:
Drug: Budesonide — budesonide starting day 5 after transplant
  Arms: Budesonide

SUMMARY:
The purpose of this study is to determine if budesonide prophylaxis starting day 5 after transplant reduces engraftment fever in autologous and allogeneic stem cell transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* • Patients 18-80 years of age with a diagnosis of a hematological malignancy

  * Meet the BMT program criteria to undergo hematopoietic stem cell transplantation for hematologi malignancies

Exclusion Criteria:

* • Patients enrolled in investigational clinical trials

  * Sct for non hematologic malignancies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
non-infectious fever | 30 days post stem cell transplant
  non infectious fever defined as fever without identified infection that occurs up to 3 days prior and 10 days after the day of engraftment in patients on budesonide prophylaxis compared to patients who will not receive prophylaxis

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States